CLINICAL TRIAL: NCT07287501
Title: Efficacy of Pain Science Education Combined With Exercise in Older Adults With Chronic Pain
Acronym: PSE-EX-OA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Javier Torres Alonso, Graduate in physiotherapy, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USalamancanº1424
Record Dates: First submitted 2025-11-18; First posted 2025-12-17 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Chronic Pain
Keywords: "Pain Education"; "Patient Education",; "Exercise"; "Healthy Aging"; "Aged"
MeSH Terms: conditions — Chronic Pain; Motor Activity | interventions — Patient Education as Topic; Exercise

STUDY DESIGN:
Intervention Model Description: An experimental, prospective, and longitudinal study was proposed. A randomized clinical trial with three groups in a 1:1:1 ratio was conducted, in which adults over 65 years of age with chronic pain were recruited.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to the nature of the intervention, it was not possible to implement complete blinding of the study participants. However, the study employed a single-blind design, in which the professionals responsible for the assessments were unaware of the participants' allocation to the intervention or control groups. Likewise, the statistical analyses were performed using coded data to ensure the objectivity of the independent researcher responsible for the statistical evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Multicomponent training control group (GC). (Active Comparator): The CG implemented a multicomponent training program lasting 32 weeks. Sessions were held three times a week, each lasting 50 minutes. The program included strength, balance, endurance, and mobility training, with individualized intensity adjustments based on progression and perceived exertion, using the Borg scale (<7) as a reference.
  Interventions: Other: Multicomponent training
- Multicomponent training group and ECD for 8 weeks (GI1). (Experimental): GI1 completed the same multicomponent training as the CG, but supplemented it with an 8-week ECD program. This training consisted of two 15-minute sessions per week (16 classes total), which addressed topics such as the difference between acute and chronic pain, neuroplasticity, the biopsychosocial approach to pain, and the impact on older adults. Supporting information was provided through presentations with images, brochures distributed at key moments, and review questionnaires, concluding with a resource and social support sheet.
  Interventions: Other: Multicomponent training combined with Pain Science Education during 8 weeks
- Multicomponent training group and ECD for 32 weeks (GI2). (Experimental): GI2 combined the same multicomponent training as CG with an extended ECD program over 32 weeks. The first 8 weeks included two 15-minute sessions per week, followed by a biweekly session, completing 24 classes. The initial content was the same as GI1, but subsequent sessions reinforced concepts through lectures, videos, role-playing, clinical case studies, and debates. Dietary guidelines, relaxation techniques, and a final guided self-reflection session were also included. The support materials included the same content as GI1, along with cards and resources specific to the dynamics.
  Interventions: Other: Multicomponent training combined with Pain Science Education during 32 weeks

INTERVENTIONS:
Other: Multicomponent training combined with Pain Science Education during 8 weeks — The intervention included multicomponent training, identical to that of the control group, combined with Pain Science Education lasting eight weeks, with two 15-minute sessions per week, totaling 16 sessions (240 minutes). The educational content covered topics such as pain, subjectivity and context, sensory homunculus and neurotag, the difference between acute and chronic pain, the distinction between damage and pain, the impact of chronic pain on older adults, the biopsychosocial approach to pain, exercise for long-term pain, attention and efferent copy, neuroplasticity, and relapses. To support the educational sessions, a PowerPoint with illustrative images and texts was used, along with two leaflets delivered at key points in the program. The first leaflet, titled "Pain Science Education," was provided at the midpoint along with an envelope to store the materials. The second leaflet, "Active Pain Coping," was given during the penultimate session. To reinforce and consolidate learni
  Other Names: Patient Education; neuroscience pain education; Pain science education; pain education
  Arms: Multicomponent training group and ECD for 8 weeks (GI1).
Other: Multicomponent training — The intervention consisted of multicomponent training lasting 32 weeks, with three 50-minute sessions per week. The training included strength, balance, endurance, and mobility exercises, with intensity adjusted according to each participant's individual progression and perceived exertion, using the Borg scale (<7) as a reference.
  Other Names: exercise; strenght exercise
  Arms: Multicomponent training control group (GC).
Other: Multicomponent training combined with Pain Science Education during 32 weeks — The intervention combined multicomponent training, identical to the control group, with a 32-week Pain Science Education program. Physical training, three 50-minute sessions per week, included strength, balance, endurance, and mobility exercises, with intensity individualized based on progression and perceived exertion (Borg <7), supervised by physiotherapists. Education consisted of 24 sessions (15 minutes each): two weekly sessions during the first eight weeks and one session every two weeks thereafter. The first 16 sessions covered foundational topics, while the remaining eight reinforced concepts through talks, videos, role playing, problem-based learning, and guided debates. Practical tools included nutrition guidance, relaxation techniques, and a final guided self-reflection. Supporting materials included presentations, leaflets, a projector, and personalized cards for interactive activities.
  Other Names: pain education; neuroscience pain education; Patient Education; Pain science education
  Arms: Multicomponent training group and ECD for 32 weeks (GI2).

SUMMARY:
As people live longer, long-term pain becomes more common in old age. This type of pain can greatly affect quality of life, reduce independence in daily activities, and diminish overall well-being.

This study is part of a project called PReGe, which aims to help older adults age actively and healthily through preventive physiotherapy. The goal is to determine whether a combination of adapted exercise and education about how pain works can help improve the lives of those who suffer from it.

The study is supported by the City Council of Salamanca and the Faculty of Nursing and Physiotherapy, and it is carried out in collaboration with the Doctoral Program in Health, Disability, Dependency, and Well-being at the University of Salamanca.

The purpose of this study is to determine whether a program that combines physical exercise with educational sessions about pain is more effective for adults over 65 years of age with chronic pain, compared to doing exercise alone. The study aims to find out whether this program improves pain, understanding of pain, mobility, quality of life and Quantitative Electroencephalography (qEEG).

This is a medical research study involving participants aged 65 years or older who have experienced pain for more than three months, with an intensity of at least 3 on a 0-to-10 scale. Participants will be randomly assigned to one of three groups, each following a different type of program:

Group 1 (Control Group): will perform only adapted physical exercise. Group 2: will perform the same physical exercise and attend educational sessions about pain for 8 weeks.

Group 3: will also perform the physical exercise and attend the educational sessions, but for a period of 32 weeks.

The study will last for one full year. The exercise program will be supervised by physiotherapists, carried out over 32 weeks, three times per week, with each session lasting approximately 50 minutes. The educational sessions on pain will be brief-about 15 minutes each-and will take place immediately before the exercise sessions.

During the first two months, there will be two educational talks per week. After the Christmas break, Group 3 will continue with one talk every two weeks until the end of the study.

Three evaluations will be conducted: one before starting the program, another at two months (questionnaires and qEEG only), and a final one at nine months. The initial and final evaluation sessions will last approximately 75 minutes per participant, while the intermediate evaluation of the questionnaires will take about 45 minutes per person.

The evaluators who conduct the assessments will not know which group each participant belongs to, to ensure that the results are as objective as possible.

DETAILED DESCRIPTION:
During the course of the study, the following information will be collected, and the following types of tests and assessments will be carried out:

Personal information and medical history.

Physical condition assessments:

1. Functional assessment: the following tests will be conducted: Short Physical Performance Battery (SPPB) and Timed Up & Go (TUG).
2. Muscle strength assessment: the following tests will be performed: handgrip strength test using a JAMAR dynamometer, five-times sit-to-stand test, and force-velocity profiling using an ADR Encoder.
3. Body composition assessment: will be obtained by bioelectrical impedance analysis (BIA), including measurements of body weight, body mass index (BMI), body fat, visceral fat, appendicular muscle mass, and appendicular mass index.

Questionnaires:

1. Numerical Rating Scale for Pain (NRS)
2. Tampa Scale for Kinesiophobia (TSK-11SV)
3. Pain Catastrophizing Scale
4. Spanish version of the Graded Chronic Pain Scale
5. SF-12 Health Survey

Quantitative Electroencephalography (qEEG): (Spectral domain (brain frequencies, absolute and relative power by band), functional connectivity indices (coherence between regions), topographical or localization indices, complexity or temporal dynamics indices).

All assessments will be administered by a trained and blinded physiotherapist under optimal hygiene and safety conditions, using certified equipment and instruments.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 65 years of age
* History of pain lasting more than 3 months.
* Pain intensity of at least 3 out of 10 on the numeric pain rating scale.
* Ability to understand, speak, and write in Spanish.

Exclusion Criteria:

* Severe cognitive impairment (score < 24 on the Mini-Mental State Exam).
* Psychiatric disorders.
* Uncontrolled systemic or inflammatory conditions.
* Uncontrolled cardiac conditions.
* Any other circumstances deemed by the investigators that could interfere with the study's purpose or conduct.

Elimination Criteria:

- Attendance below 85% of total sessions.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Scale (NRS) | 32 weeks
  The Numeric Rating Scale (NRS) is a one-dimensional tool used to measure the intensity of pain perceived by an individual at a given time. It is based on self-assessment by the patient, who assigns a numerical value from 0 to 10 to their pain, where 0 indicates total absence of pain and 10 represents the worst pain imaginable. Pain between 1 and 3 is considered mild pain, between 4 and 7 moderate, and 8 to 10 severe. This variable is classified as a continuous quantitative variable. The NRS is administered in written form, is easy to understand, and does not require complex instruments, allowing its use in various clinical settings. It has been shown to be feasible and to show high correlations with other pain assessment tools. Furthermore, it is suitable for older adults with chronic pain participating in interdisciplinary pain rehabilitation.

SECONDARY OUTCOMES:
Tampa Scale for Kinesiophobia (TSK-11) | 32 weeks
  The TSK-11 is a shortened self-report tool used to assess fear of movement. It consists of 11 items scored on a 4-point Likert scale (1 = strongly disagree to 4 = strongly agree), with a total score ranging from 11 to 44, where higher scores indicate greater levels of kinesiophobia. The TSK-11 was developed as a reduced version of the original 17-item scale after psychometric analysis identified six items with low statistical performance. Studies have shown that the TSK-11 has adequate internal consistency (Cronbach's alpha = 0.79), good test-retest reliability (ICC = 0.81; SEM = 2.54), as well as concurrent and predictive validity comparable to the original scale. It also demonstrated responsiveness to change (SRM = -1.11), making it suitable for evaluating therapeutic progress. This variable is considered continuous quantitative and is particularly relevant in research addressing psychosocial factors related to chronic pain and functional disability.
Pain Catastrophizing Scale (PCS) | 32 weeks
  A 13-item self-report tool assessing negative thoughts about pain across rumination, magnification, and helplessness. Each item is scored 0-4 (total 0-52); higher scores indicate greater catastrophizing. It is reliable, valid, and important in chronic pain management.
Graded Chronic Pain Scale (GCPS) | 32 weeks
  An 8-item scale measuring pain intensity and disability (total 0-70). Quick to administer, reliable, valid, and useful for classifying pain severity and functional impact.
SF-12 Health Survey | 32 weeks
  A 12-item questionnaire assessing physical and mental health-related quality of life. Produces standardized scores and is widely used in research and clinical practice.
Sociodemographic Variables | 32 weeks
  For each patient, the following data were recorded: full name, ID number, phone number, sex, marital status, medical history, presence of chronic conditions (such as hypertension, diabetes, high cholesterol, hypothyroidism, among others), use of additional medications, number of tablets taken daily, number of analgesics taken daily, living situation, educational level, and general clinical condition. Blood pressure and heart rate were also measured to ensure that the patient was in optimal condition to undergo the evaluations.
Short Physical Performance Battery (SPPB) | 32 weeks
  A widely used tool in geriatric research to assess physical performance. It includes three tests measuring lower limb strength, gait speed, and balance. Total scores range from 0 to 12, with up to 4 points per component. Scores below 8 indicate low physical performance. The SPPB is quick, requires minimal equipment, and has high test-retest reliability, predictive validity, and clinical applicability.
Timed Up & Go (TUG) | 32 weeks
  Assesses mobility and balance by timing how long a person takes to stand from a chair, walk 3 meters, turn, return, and sit down. The test is performed twice, taking the best time. Times exceeding age-specific thresholds indicate below-average performance: >9.0s (60-69 years), >10.2s (70-79 years), >12.7s (80-99 years).
Handgrip strength (JAMAR dynamometer) | 32 weeks
  Measures grip strength quantitatively in kilograms. Performed seated with elbow at 90º and neutral hand position. Each hand is tested alternately, taking the average. The JAMAR dynamometer shows excellent reproducibility and interrater reliability and is considered the gold standard for handgrip assessment.
Force-velocity profile (ADR Encoder) | 32 weeks
  Evaluates the relationship between muscle force and contraction speed. Measured during five rapid sit-to-stand repetitions using a linear encoder attached at the waist, recording power, speed, and distance. Reliable in older adults and useful for performance optimization.
Body Mass Index (BMI) | 32 weeks
  Weight (kg) divided by height (m²). Classifies individuals into ranges and serves as a screening tool for body composition and risk of chronic disease, though it does not directly measure fat percentage.
Body fat percentage | 32 weeks
  Indicates proportion of fat relative to total body weight. Normal ranges: men 12-20%, women 24-30%; obesity: men >25%, women >33%. Distribution (visceral vs. subcutaneous) is important for disease risk.
Visceral fat | 32 weeks
  Fat surrounding internal organs, ~10% of total body fat, linked to higher risk of cardiovascular, metabolic, and other diseases.
Appendicular skeletal muscle mass (ASM) | 32 weeks
  Muscle mass in arms and legs. Measured via BIA, DXA, MRI, or anthropometry. BIA provides validated estimations of lean mass over time.
Skeletal Muscle Index (SMI) | 32 weeks
  ASM adjusted for height (ASM/height²) to account for body size, as recommended by EWGSOP2.
Abdominal circumference | 32 weeks
  Measured at the navel after full exhalation. Values >102 cm in men and >88 cm in women indicate increased health risk, providing information independent of BMI on central adiposity.
Change in Resting State Absolute Power of the Alpha Band | 32 weeks
  Quantitative Electroencephalography (qEEG) will be used to assess cortical activity. The signal will be decomposed using Fast Fourier Transform (FFT). The specific outcome is the mean absolute power in the Alpha frequency band (8-12 Hz) across the regions of interest (ROIs). Changes in alpha power are associated with pain modulation and central sensitization mechanisms. Unit of Measure:
  Microvolts squared
Change in Functional Connectivity (Inter-regional Coherence) | 32 weeks
  Functional connectivity between brain regions will be assessed using spectral coherence indices derived from the qEEG. Coherence indicates the degree of synchronization between two brain regions at specific frequencies. Values range from 0 (no correlation) to 1 (perfect correlation). This metric evaluates the integration of neural networks involved in pain processing. Unit of Measure: Coherence coefficient (0-1)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing and Physiotherapy USAL. Campus Miguel de Unamuno, C. Donantes de Sangre, s/n, 37007 Salamanca, Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Yes
The anonymized Individual Participant Data (IPD) set supporting the main publication will be made available to other researchers. This will include data from the Quantitative Electroencephalography (qEEG) variables, behavioral measures, and relevant demographic variables, always ensuring the non-identification of participants, as established in the approved informed consent. Data will be accessible starting 6 months after the primary article's publication, with no end date. Access will be granted upon formal request to the Principal Investigator, submission of a methodologically sound research proposal, and the signing of a Data Use Agreement (DUA) to ensure the protection of participant privacy.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The data and supporting information (Study Protocol, Statistical Analysis Plan, Informed Consent Form, and Analytical Code) will be available starting 6 months after the publication of the main manuscript in a scientific journal, and will remain available indefinitely through the Principal Investigator or a permanent data repository.
Access Criteria: Access to the anonymized IPD and supporting documents (Protocol, SAP, ICF, Analytical Code) is granted to qualified scientific investigators whose proposal is deemed methodologically sound and aligns with the study's ethical goals. Requests must be submitted formally to the Principal Investigator. Access requires the applicant to sign a Data Use Agreement (DUA), ensuring compliance with the confidentiality measures set forth in the original informed consent, and adherence to relevant data protection regulations (e.g., GDPR). The DUA will strictly prohibit any attempt at participant re-identification and must include a commitment to using the data solely for the approved research purpose.

REFERENCES:
- [Background] Soares Fonseca L, Pereira Silva J, Bastos Souza M, Gabrich Moraes Campos M, de Oliveira Mascarenhas R, de Jesus Silva H, Souza Maximo Pereira L, Xavier Oliveira M, Cunha Oliveira V. Effectiveness of pharmacological and non-pharmacological therapy on pain intensity and disability in older people with chronic nonspecific low back pain: a systematic review with meta-analysis. Eur Spine J. 2023 Sep;32(9):3245-3271. doi: 10.1007/s00586-023-07857-4. Epub 2023 Jul 18. PMID 37464184
- [Background] Lam N, Green J, Hallas S, Forster A, Crocker TF, Andre D, Ellwood A, Clegg A, Brown L. Mapping review of pain management programmes and psychological therapies for community-dwelling older people living with pain. Eur Geriatr Med. 2024 Feb;15(1):33-45. doi: 10.1007/s41999-023-00871-1. Epub 2023 Oct 18. PMID 37853269
- [Background] Zahari Z, Ishak A, Justine M. The effectiveness of patient education in improving pain, disability and quality of life among older people with low back pain: A systematic review. J Back Musculoskelet Rehabil. 2020;33(2):245-254. doi: 10.3233/BMR-181305. PMID 31356191
- [Background] Watson JA, Ryan CG, Atkinson G, Williamson P, Ellington D, Whittle R, Dixon J, Martin DJ. Inter-Individual Differences in the Responses to Pain Neuroscience Education in Adults With Chronic Musculoskeletal Pain: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Pain. 2021 Jan;22(1):9-20. doi: 10.1016/j.jpain.2020.03.006. Epub 2020 Jun 22. PMID 32585363
- [Background] Nunez-Cortes R, Salazar-Mendez J, Calatayud J, Malfliet A, Lluch E, Mendez-Rebolledo G, Guzman-Munoz E, Lopez-Bueno R, Suso-Marti L. The optimal dose of pain neuroscience education added to an exercise programme for patients with chronic spinal pain: a systematic review and dose-response meta-analysis. Pain. 2024 Jun 1;165(6):1196-1206. doi: 10.1097/j.pain.0000000000003126. Epub 2023 Nov 30. PMID 38047772
- [Background] Nijs J, Paul van Wilgen C, Van Oosterwijck J, van Ittersum M, Meeus M. How to explain central sensitization to patients with 'unexplained' chronic musculoskeletal pain: practice guidelines. Man Ther. 2011 Oct;16(5):413-8. doi: 10.1016/j.math.2011.04.005. Epub 2011 May 31. PMID 21632273
- [Background] Sluka KA, Frey-Law L, Hoeger Bement M. Exercise-induced pain and analgesia? Underlying mechanisms and clinical translation. Pain. 2018 Sep;159 Suppl 1(Suppl 1):S91-S97. doi: 10.1097/j.pain.0000000000001235. PMID 30113953
- [Background] Carville S, Constanti M, Kosky N, Stannard C, Wilkinson C; Guideline Committee. Chronic pain (primary and secondary) in over 16s: summary of NICE guidance. BMJ. 2021 Apr 21;373:n895. doi: 10.1136/bmj.n895. No abstract available. PMID 33883123
- [Background] Castellini G, Iannicelli V, Briguglio M, Corbetta D, Sconfienza LM, Banfi G, Gianola S. Are clinical practice guidelines for low back pain interventions of high quality and updated? A systematic review using the AGREE II instrument. BMC Health Serv Res. 2020 Oct 22;20(1):970. doi: 10.1186/s12913-020-05827-w. PMID 33092579
- [Background] Cai Y, Leveille SG, Shi L, Chen P, You T. Chronic pain and circumstances of falls in community-living older adults: an exploratory study. Age Ageing. 2022 Jan 6;51(1):afab261. doi: 10.1093/ageing/afab261. PMID 35061871
- [Background] Lin T, Zhao Y, Xia X, Ge N, Yue J. Association between frailty and chronic pain among older adults: a systematic review and meta-analysis. Eur Geriatr Med. 2020 Dec;11(6):945-959. doi: 10.1007/s41999-020-00382-3. Epub 2020 Aug 17. PMID 32808241
- [Background] Domenichiello AF, Ramsden CE. The silent epidemic of chronic pain in older adults. Prog Neuropsychopharmacol Biol Psychiatry. 2019 Jul 13;93:284-290. doi: 10.1016/j.pnpbp.2019.04.006. Epub 2019 Apr 17. PMID 31004724
- [Background] Cimas M, Ayala A, Sanz B, Agullo-Tomas MS, Escobar A, Forjaz MJ. Chronic musculoskeletal pain in European older adults: Cross-national and gender differences. Eur J Pain. 2018 Feb;22(2):333-345. doi: 10.1002/ejp.1123. Epub 2017 Dec 12. PMID 29235193
- See also: World Population Prospects [Internet]. [cited 2025 Apr 2]. — https://population.un.org/wpp/downloads?folder=Standard%20Projections&group=Most%20used